CLINICAL TRIAL: NCT03099213
Title: A Study of Patients Treated With Ramipril for Cardiovascular Risk Reduction The HOPE Tips: The HOPE Study Translated Into PracticeS
Brief Title: An Open-label, Non-comparative Study to Document the Tolerability to Ramipril in Patients With at Least One High Risk for Developing a Major Cardiovascular Event
Acronym: HOPETips
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAMIP_L_03123; U1111-1193-0859 (Other: UTN)
Record Dates: First submitted 2017-03-31; First posted 2017-04-04 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramipril (Experimental): Receiving ramipril with the recommended initial dose of 2.5 mg once daily; depending on the tolerability, the dose should be gradually increased. The increase should be implemented by doubling the dose after one to two weeks. Three or four weeks later, the dose should be doubled again up to the usual maintenance dose of 10 mg once daily.
  Interventions: Drug: RAMIPRIL HOE498

INTERVENTIONS:
Drug: RAMIPRIL HOE498 — Pharmaceutical form:Tablet Route of administration: Oral

SUMMARY:
Primary Objective:

To document the tolerability of patients receiving study medication at 12-week of therapy in terms of the scoring system assessed by the investigator.

Secondary Objectives:

* To document drug safety at 12-week of treatment in terms of number of Adverse Drug Reaction or Serious Adverse Drug Reaction reported.
* To describe the population treated as per the HOPE study indication in current clinical practice (demographics, cardiovascular risk-factors at treatment initiation, concomitant treatments patterns).

DETAILED DESCRIPTION:
The duration of the study period is 8-12 weeks.

ELIGIBILITY:
Inclusion criteria :

* Man or woman, age 55 years old or more.
* Presence of a high risk of developing a major cardiovascular event, defined as at least one of the following underlying conditions:
* Clinical evidence of coronary artery disease (examples: previous myocardial infarction [MI], positive stress test or significant stenosis at coronary angiography, previous Percutaneous Trans-Luminal Coronary Angioplasty [PTCA], previous Coronary Arterial Bypass Grafting [CABG]);
* Clinical evidence of peripheral vascular disease (examples: history of intermittent claudication with positive Doppler or angiography, previous limb bypass surgery, previous percutaneous trans-luminal angioplasty, previous limb or foot amputation);
* Previous stroke;
* Diabetes (insulin-dependent or non-insulin dependent) with at least one of the following cardiovascular risk factors:
* hypertension (blood pressure [BP] >140/90 mmHg, or patients on antihypertensive treatment);
* hypercholesterolemia (total cholesterol > 5.2 mmol/L [>200 mg/dL]);
* low HDL cholesterol (< 0.9 mmol/L [<3.5 mg/dL]);
* current cigarette smoking;
* documented microalbuminuria (30-300 mg/24 hours);
* Evidence of previous vascular disease.

Exclusion criteria:

* Patients with contraindications to ramipril use (as per the local Ramipril Product Information)
* hypersensitivity
* pregnancy, lactation
* bilateral renal stenosis
* Patients with clinically relevant concomitant disease that could compromise the patient's safety or follow up.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2008-11-01; Primary Completion 2010-04-23 (Actual); Study Completion 2010-04-23 (Actual)

PRIMARY OUTCOMES:
Total patients with tolerability score Very Good | 12 weeks
Total patients with tolerability score Good | 12 weeks
Total patients with tolerability score Sufficient | 12 weeks
Total patients with tolerability score Insufficient | 12 weeks
Total patients with tolerability score Not Good | 12 weeks

SECONDARY OUTCOMES:
Number of Adverse Events or Serious Adverse Events reported | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi Administrative Office, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org